CLINICAL TRIAL: NCT03527329
Title: Perioperative Hypothermia in Patients Submitted to Transurethral Resection
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Ángel Becerra, MD, Dr. Negrin University Hospital
Other Study IDs: NAC120300
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Hypothermia; Anesthesia; Peroperative Complication
Keywords: Prewarming; Tympanic temperature
MeSH Terms: conditions — Hypothermia; Intraoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prewarming: Active Prewarming will be performed using a forced-air blanket (WarmTouch lower body blanket, Covidien Ltd, Mansfield, USA) over the whole body and connected to a forced-air warmer (WarmTouch Model 5900, Covidien Ltd, Mansfield, USA). Patients will be warmed using a surgical blanket during the intraoperative period. Tympanic thermometer (Genius 2 Tympanic Thermometer and Base, Covidien Ltd, Mansfield, USA) will be used to measure the temperature throughout the perioperative period.
  Interventions: Device: WarmTouch Model 5900, Covidien Ltd, Mansfield, USA
- Control: Non-active prewarming. Patients will be warmed using a surgical blanket during the intraoperative period. Tympanic thermometer (Genius 2 Tympanic Thermometer and Base, Covidien Ltd, Mansfield, USA) will be used to measure the temperature throughout the perioperative period.

INTERVENTIONS:
Device: WarmTouch Model 5900, Covidien Ltd, Mansfield, USA — Forced-air warming will be applied following routine clinical practice. The pre-warming time will depend on the time the patient has to wait before entering in the operating room. Prewarming time will be recorded for each patient.
  Groups: Prewarming

SUMMARY:
Hypothermia is a frequent perioperative complication. Its appearance can have deleterious effects such as myocardial ischemia or perioperative bleeding. When the negative effects of anesthesia on temperature are aggravated by other factors, such as glycine infusion in transurethral resection, temperature can decrease even more. Once the temperature has decreased, its treatment is difficult. Preoperative warming prevents hypothermia, lowering the temperature gradient between core and peripheral compartments and reducing thermal redistribution. The most recent clinical practice guidelines advocate for active prewarming before induction of general anaesthesia since it is very effective in preventing perioperative hypothermia. However, the ideal warming time prior to the induction of anesthesia has long been investigated. This study aims to evaluate if different time periods of preoperative forced-air warming reduces the incidence of hypothermia at the end of surgery in patients submitted to transurethral resection. This is an observational prospective study comparing routine practice of pre-warming in consecutive surgical patients scheduled to undergo elective transurethral resection between March 2014 and April 2018. Three-hundred patients are included in this study and prewarming will be applied following routine clinical practice. The prewarming time will depend on the time the patient has to wait before entering in the operating theatre. Measurement of temperature will be performed using a tympanic thermometer. Patients will be followed throughout their hospital admission. Data will be recorded using a validated instrument and will be analysed using the statistics program R Core Team.

DETAILED DESCRIPTION:
Maintaining patient's temperature above 36 grades Celsius throughout the perioperative period is challenging. Thus, it is essential to monitor temperature in order to be able to take measures to avoid the appearance of hypothermia. Once the temperature has decreased, its treatment is difficult since the application of heat to the body surface takes a long time to reach the core thermal compartment. Intraoperative warming alone cannot avoid postoperative hypothermia. The application of forced-air warming system during the preoperative period has been shown to be the most effective measure to prevent hypothermia and maintain intraoperative normothermia. However, it would not be efficient to provide a long-time prewarming in short-term surgical procedures. Thus, the ideal warming time prior to the induction of anesthesia has long been investigated.

Due to the searching of optimal prewarming time and the lack of evidence about the efficiency of prewarming in patients submitted to transurethral resection, the conductance of this study is justified.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective Transurethral resection under general or spinal anesthesia.

Exclusion Criteria:

* Active infection
* Intake of antipyretics within 24 hours before surgery
* Neuropathy
* Thyroid disorders
* Peripheral vascular disease
* Skin lesions
* History of hypersensitivity to skin contact devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an observational prospective study comparing routine practice of pre-warming in consecutive surgical patients scheduled to undergo elective transurethral resection between March 2014 and April 2018. Three-hundred patients are included in this study and prewarming will be applied following routine clinical practice. The prewarming time will not be decided by the clinical investigator. Prewarming time will depend on the time the patient has to wait before entering in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Temperature | Through patient's stay in hospital, an average of 24 hours
  Asses the effect of prewarming in maintaining body temperature of patients undergoing elective transurethral resection.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelio Rodríguez-Pérez, MD PhD, Study Director — Dr. Negrin University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] NICE. Inadvertent Perioperative Hypothermia: The Management of Inadvertent Perioperative Hypothermia in Adults. NICE Clinical Guideline No. 65, 2008.
- [Background] Hooper VD, Chard R, Clifford T, Fetzer S, Fossum S, Godden B, Martinez EA, Noble KA, O'Brien D, Odom-Forren J, Peterson C, Ross J, Wilson L; ASPAN. ASPAN's evidence-based clinical practice guideline for the promotion of perioperative normothermia: second edition. J Perianesth Nurs. 2010 Dec;25(6):346-65. doi: 10.1016/j.jopan.2010.10.006. No abstract available. PMID 21126665
- [Background] Torossian A, Brauer A, Hocker J, Bein B, Wulf H, Horn EP. Preventing inadvertent perioperative hypothermia. Dtsch Arztebl Int. 2015 Mar 6;112(10):166-72. doi: 10.3238/arztebl.2015.0166. PMID 25837741
- [Background] Forbes SS, Eskicioglu C, Nathens AB, Fenech DS, Laflamme C, McLean RF, McLeod RS; Best Practice in General Surgery Committee, University of Toronto. Evidence-based guidelines for prevention of perioperative hypothermia. J Am Coll Surg. 2009 Oct;209(4):492-503.e1. doi: 10.1016/j.jamcollsurg.2009.07.002. Epub 2009 Aug 20. No abstract available. PMID 19801323